CLINICAL TRIAL: NCT00140712
Title: A Study to Determine the Tolerability and Pharmacokinetics for Ropinirole in Paediatric / Adolescent Patients With RLS (Type 2)
Brief Title: Ropinirole Tablets In Young Patients With Restless Legs Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101468/253
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Restless Legs Syndrome
Keywords: RLS; PLMS; Adolescent; Periodic Limb Movements of Sleep; Ropinirole
MeSH Terms: conditions — Restless Legs Syndrome | interventions — ropinirole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ropinirole (Experimental): single dose .25mg of IR formulation, .05mg of RLS controlled release
  Interventions: Drug: Ropinirole Immediate Release

INTERVENTIONS:
Drug: Ropinirole Immediate Release — Ropinirole Immediate Release

SUMMARY:
This is a two-period dose rising study of Ropinirole Immediate Release in adolescent patients with restless legs syndrome (RLS) in order to determine the starting dose for the ropinirole titration regimen for this age group. Patients will receive two single doses unless poor tolerability is observed following the first dose.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent subjects diagnosed with probable or definite Restless Leg Syndrome (RLS).

Exclusion Criteria:

* Subjects who require RLS treatment during the daytime, suffer from other primary sleep disorders or are taking medication known to induce drowsiness, affect RLS or sleep, or to induce or treat alertness, including methylphenidate.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2005-06-10 (Actual); Primary Completion 2008-02-28 (Actual); Study Completion 2008-02-28 (Actual)

PRIMARY OUTCOMES:
AUC(0-8), Cmax. Safety (adverse events, vital signs, ECG, laboratory parameters), Change in BP, Incidence of adverse events. Number of periodic limb movements and Number of periodic limb movements per hour (as measured by actigraphy). | Up to 3 years

SECONDARY OUTCOMES:
PK - tmax, t1/2, For SKF-89124 and SKF-104557 - ratio of metabolite AUC:ropinirole AUC. PD - Leg movement as measured by actigraphy. | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- United States (7):
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, Chapel Hill, North Carolina
- GSK Investigational Site, Brussels, Belgium
- GSK Investigational Site, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 101468/253 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/101468/253?search=study&study_ids=101468%2F253#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 101468/253 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 101468/253 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 101468/253 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 101468/253 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 101468/253 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 101468/253 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 101468/253 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register